CLINICAL TRIAL: NCT02018575
Title: Application of the Indicator Amino Acid Oxidation Technique for the Determination of Metabolic Availability of Lysine From White Maize Protein, in Young Adult Men
Brief Title: Metabolic Availability of Lysine From White Maize
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Dr. Paul Pencharz, Professor of Paediatrics and Nutritional Sciences (Emeritus) University of Toronto, Senior Scientist Research Institute, The Hospital for Sick Children, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0019850580 amendment
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Adults
Keywords: lysine; bioavailability; amino acids; corn
MeSH Terms: conditions — Callosities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- levels of lysine intake. (Experimental): Randomly selected levels of lysine intake which are lower than the lysine requirement (previously derived).
  Interventions: Dietary Supplement: Crystalline Lysine Amino Acid Mix; Dietary Supplement: White corn meal porridge

INTERVENTIONS:
Dietary Supplement: Crystalline Lysine Amino Acid Mix — Crystalline Lysine from Amino Acid Mixture in amount of 29, 37, 46 and 54% of the mean Lysine requirement of 35 mg/kg/d will be given to subjects.
Dietary Supplement: White corn meal porridge — A cornmeal porridge including 29, 37, 46 and 54% of the mean Lysine requirement of 35 mg/kg/d will be given to subjects.

SUMMARY:
Our objective is to determine the metabolic availability of Lysine in white maize using the indicator amino acid oxidation (IAAO) technique in adult men.

DETAILED DESCRIPTION:
Our objective is to determine the metabolic availability of Lysine in white maize. 7 young, healthy, male adults will receive graded levels (29, 37,46 and 54%) of lysine requirement of 35 mg/kg/d as a crystalline AA mixture and a porridge of white cornmeal protein respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult males (20-49 years old)

Exclusion Criteria:

* A history of recent weight loss or illness
* Use of any medication at the time of entry into the study

Ages: 20 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2013-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Metabolic Availability of Lysine | Baseline
  3 breath samples will be taken to provide a baseline F13CO2 measurement (Level of Phenylalanine oxidation). Breath samples will be collected and analyzed for 13CO2 enrichment.

SECONDARY OUTCOMES:
Metabolic Availability of Lysine | 15 mins after intake of the fourth hourly meal (before tracer infusion)
  3 breath samples will be taken to provide a baseline F13CO2 measurement (Level of Phenylalanine oxidation). Breath samples will be collected and analyzed for 13CO2 enrichment.

OTHER OUTCOMES:
Metabolic availability of Lysine | 30 mins after intake of the fourth hourly meal (before tracer infusion)
  3 breath samples will be taken to provide a baseline F13CO2 measurement (Level of Phenylalanine oxidation). Breath samples will be collected and analyzed for 13CO2 enrichment.
Metabolic Availability of Lysine | 45 mins after intake of the fourth hourly meal (before tracer infusion)
  3 breath samples will be taken to provide a baseline F13CO2 measurement (Level of Phenylalanine oxidation). Breath samples will be collected and analyzed for 13CO2 enrichment.
Metabolic Availability of Lysine | Post Tracer Infusion (between 150 and 240 min of tracer infusion)
  4 breath samples will be taken to provide F13CO2 measurement (Level of Phenylalanine oxidation). Breath samples will be collected and analyzed for 13CO2 enrichment.

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Pencharz, MD, PhD, Principal Investigator — The Hospital for Sick Children, Toronto, Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada